CLINICAL TRIAL: NCT00648596
Title: An International, Multicentre, Randomized, Parallel Group, Double Blind, Placebo Controlled, Flexible Dose Study to Evaluate Self-esteem and Relationships in Males With Erectile Dysfunction Treated With Sildenafil Citrate
Brief Title: A Study to Evaluate Self-esteem and Relationships in Males With Erectile Dysfuntion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1481161
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 2 (Placebo Comparator)
  Interventions: Drug: placebo
- Arm 1 (Active Comparator)
  Interventions: Drug: sildenafil

INTERVENTIONS:
Drug: sildenafil — sildenafil 50 mg tablet by mouth 1 hour before sexual activity for 12 weeks; the dose could be increased to 100 mg or decreased to 25 mg.
  Arms: Arm 1
Drug: placebo — placebo tablet by mouth 1 hour before sexual activity for 12 weeks
  Arms: Arm 2

SUMMARY:
To determine the improvement in the self-esteem domain score of the Self-Esteem/Overall Relationship (SEAR) questionnaire and the improvement in erectile function (obtained from the Erectile Function [EF] domain of the International Index of Erectile Function [IIEF]). Furthermore, to determine if the improvement obtained in self-esteem was related to the main erectile dysfunction (ED) co-morbidities type and/or number.

ELIGIBILITY:
Inclusion Criteria:

-Men with a documented clinical diagnosis of ED confirmed by a Sexual Health Inventory-Male (SHI-M) score of 21 or less and who have a sexual partner for the duration of the study were included.

Exclusion Criteria:

* Subjects who have previously taken, or it is suspected they have taken, more than 4 doses of sildenafil citrate, or any other phosphodiesterase type 5 (PDE-5) inhibitor, or apomorphine, at any time prior to the screening visit or patients who have taken any dose of these compounds in the last two months
* Subjects with resting sitting hypotension (BP < 90/50mmHg) or hypertension (BP > 170/110mmHg)
* Subjects with significant cardiovascular disease, including cardiac failure, myocardial infarction, unstable angina, stroke or transient ischaemic attack (TIA), symptomatic or clinically significant cardiac arrhythmias in the last 3 months
* Patients on nitrates.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Actual)
Dates: Start 2003-05; Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Self-esteem domain of the SEAR questionnaire | Week 12

SECONDARY OUTCOMES:
Correlation between the change in the SE domain of the SEAR questionnaire and the erectile function domain of the IIEF by number of ED co-morbidities | Week 12
Differences in the global efficacy assessment question overall and by type of co-morbidity | Week 12
Differences in the global satisfaction assessment questions overall and by type of co-morbidity | Week 12
Comparisons between treatments in the SE domain of the SEAR questionnaire by type of co-morbidity (hypertension, hyperlipidemia, diabetes mellitus, benign prostatic hyperplasia, depression) | Week 12
Changes in the sexual activity domain of the SEAR questionnaire overall and by type of co-morbidity | Week 12
Changes in the relationship domain of the SEAR questionnaire overall and by type of co-morbidity | Week 12
Changes of the SEAR questions overall and by type of co-morbidity | Week 12
Changes of the IIEF questions overall and by type of co-morbidity | Week 12
Changes of the IIEF domains overall and by type of co-morbidity | Week 12
Degrees of severity in the IIEF erectile function | Week 12
Correlation between the change in the SE domain of the SEAR questionnaire and the erectile function domain of the IIEF overall and by type of co-morbidity | Week 12
Changes in the questions from the event log overall and by type of co-morbidity | Week 12
Correlation between each success rate derived from the event log and the change in the SE domain of the SEAR questionnaire overall and by type of co-morbidity | Week 12
Differences in the intercourse success rates derived from the event log overall and by type of comorbidity | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (53):
- Finland (3):
  - Pfizer Investigational Site, Oulu
  - Pfizer Investigational Site, Tampere
  - Pfizer Investigational Site, Turku
- France (8):
  - Pfizer Investigational Site, Clermont-Ferrand
  - Pfizer Investigational Site, LE Kremlin Bicentre
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Neuilly-sur-Seine
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Nîmes
  - Pfizer Investigational Site, Toulouse
- Italy (8):
  - Pfizer Investigational Site, Bari
  - Pfizer Investigational Site, Catania
  - Pfizer Investigational Site, Gallarate (VA)
  - Pfizer Investigational Site, Modena
  - Pfizer Investigational Site, Padua
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Siena
  - Pfizer Investigational Site, Torino
- Poland (6):
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Lublin
  - Pfizer Investigational Site, Olsztyn
  - Pfizer Investigational Site, Szczecin
  - Pfizer Investigational Site, Warsaw
- Russia (7):
  - Pfizer Investigational Site, Barnaul
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Nizhny Novgorod
  - Pfizer Investigational Site, Novosibirsk
  - Pfizer Investigational Site, Rostov-on-Don
  - Pfizer Investigational Site, Saint Petersburg
  - Pfizer Investigational Site, Yekaterinburg
- Spain (6):
  - Pfizer Investigational Site, San Juan, Alicante
  - Pfizer Investigational Site, Barakaldo, Vizcaya
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Valencia
  - Pfizer Investigational Site, Zaragoza
- Sweden (6):
  - Pfizer Investigational Site, Karlshamn
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Skövde
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Värnamo
  - Pfizer Investigational Site, Västervik
- United Kingdom (9):
  - Pfizer Investigational Site, Bodelwyddan, Denbighshire
  - Pfizer Investigational Site, South Yorkshire, DN1 2ET
  - Pfizer Investigational Site, Belmont, Durham
  - Pfizer Investigational Site, Blackpool, Lancashire
  - Pfizer Investigational Site, Urmston, Manchester
  - Pfizer Investigational Site, Ashford, Middlesex
  - Pfizer Investigational Site, Nr Lichfield, Staffordshire
  - Pfizer Investigational Site, Addlestone, Surrey
  - Pfizer Investigational Site, Taunton, TA1 5DA

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481161&StudyName=An%20international%2C%20multicentre%2C%20randomized%2C%20parallel%20group%2C%20double%20blind%2C%20placebo%20controlled%2C%20flexible%20dose%20study%20to%20evaluate%20self-es